CLINICAL TRIAL: NCT04988737
Title: Usability of a Perioperative Medication-Related Clinical Decision Support Application: A Randomized Controlled Trial
Brief Title: Usability of a Perioperative Medication-Related Clinical Decision Support Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen C. Nanji,M.D.,M.P.H., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020P000210
Record Dates: First submitted 2021-07-09; First posted 2021-08-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2021-07

CONDITIONS: Perioperative Medication Errors; Perioperative Adverse Medication Events
Keywords: Usability; Clinical Decision Support; Anesthesiology; Medication Safety

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDS Group (Experimental): Clinicians complete tasks using the CDS prototype. Briefly, the clinician scans the barcode on the syringe label immediately prior to medication administration. The scan triggers the CDS to display a dosing window with pertinent patient-specific information and/or alert(s) when necessary to prevent a medication error (ME) prior to the medication being administered. Medication data are then sent from the CDS application to the patient's anesthesia record for automatic documentation in real-time, eliminating the need to manually document the medication in the Anesthesia Information Management System (AIMS). When necessary, the CDS application generates alerts to prevent medication errors. Upon receiving an alert, the anesthesia clinician may accept the alert and revise the action that generated the alert, or override the alert and continue with the planned action.
  Interventions: Other: Electronic Clinical Decision Support Application
- Control Group (No Intervention): Clinicians complete tasks using the conventional medication administration and documentation workflow in anesthesia.

INTERVENTIONS:
Other: Electronic Clinical Decision Support Application — Robust, real-time medication-related clinical decision support application for use in the operating room. The application is fully integrated with existing clinical systems. It provides visual alerts for medication errors and adverse medication events at the point-of-care.
  Arms: CDS Group

SUMMARY:
The goal of this study is to compare the usability of a novel, medication-related clinical decision support (CDS) application to the current standard medication administration and documentation workflow. The study will occur in a simulation setting, using a manikin and test patient data - no actual patients will participate. Forty clinician participants will be randomly assigned to either the CDS group (who will complete simulation tasks using the CDS prototype) or the Control group (who will complete simulation tasks using the standard medication administration workflow).

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia Clinicians including attending anesthesiologists, Certified Registered Nurse Anesthetists (CRNAs), and house staff (residents and fellows)

Exclusion Criteria:

* Study Staff
* Medical Students

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Total time to complete 7 simulations tasks. | Measured from task start time to task end time, a cumulative average of 15 minutes
  Total time (in seconds) to complete 7 simulations tasks.

SECONDARY OUTCOMES:
Total number of mouse clicks in 7 simulations tasks. | Measured from task start time to task end time, a cumulative average of 15 minutes
  Total count of mouse clicks during all 7 simulations tasks.
Total distance traveled on the screen in pixels for 7 simulation tasks. | Measured from task start time to task end time, a cumulative average of 15 minutes
  Total distance traveled on the screen in pixels during all 7 simulation tasks.

OTHER OUTCOMES:
System Usability Scale (SUS) score. | Measured at the conclusion of study participation, an average of 15 minutes after the participant's start time
  SUS is designed and validated only for first-time system users, so it will be completed by the CDS group only. SUS scores range from 0 to 100 (higher score indicates higher usability). The scores are not percentiles, but are interpreted using benchmark comparisons to industry standards.
Number of usability issues. | Identified continuously over the duration of study participation, a cumulative average of 15 mins
  Usability issues are defined as aspects of the system that prevent the user from accomplishing their goals with effectiveness, efficiency and satisfaction. Usability issues will be identified for the CDS group only. Usability issues will be identified by a usability expert.
Single Ease Question score for each simulation task. | Measured at the end of each of the 7 tasks (each task requires an average of 3 minutes to complete)
  "Overall, how difficult or easy did you find this task?" Answers will be recorded on a 7-point Likert scale (1= "very difficult"; 7= "very easy").

CONTACTS AND LOCATIONS:
Overall Officials: Karen C Nanji, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No